CLINICAL TRIAL: NCT00005218
Title: Epidemiological Tool To Detect Angina Pectoris in Blacks
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1097; R43HL040730 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2002-04

CONDITIONS: Cardiovascular Diseases; Angina Pectoris; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Angina Pectoris; Heart Diseases

SUMMARY:
To develop a prototype questionnaire for the detection of angina pectoris in Blacks.

DETAILED DESCRIPTION:
BACKGROUND:

Angina pectoris is often considered a manifestation of coronary artery atherosclerosis that is associated with an increased mortality risk. Overall, coronary heart disease is the leading cause of morbidity and mortality in United States Blacks. In an attempt to standardize the diagnosis of angina pectoris in epidemiologic studies, Rose developed a questionnaire for cardiovascular field surveys which has primarily been used in United States and other white populations. However, in 1988, there were no valid epidemiological tools for the assessment of angina pectoris in Blacks. The development of a cardiovascular survey instrument capable of assessing angina pectoris in Black populations was identified by the Association of Black Cardiologists as an urgent epidemiologic need. Also, such a survey instrument could ultimately enhance knowledge and treatment of cardiovascular disease among Blacks.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1988-04; Study Completion 1990-03 (Actual)

REFERENCES:
- [Background] Clark LT, Adams-Campbell LL, Maw M, Bridges D, Kline G. Atypical myocardial infarction and hypertension: an inner city experience. J Hum Hypertens. 1990 Apr;4(2):105-7. PMID 2338676